CLINICAL TRIAL: NCT03879551
Title: The Effect of High Frequency Repetitive Transcranial Magnetic Stimulation on Cognitive Impairment in Parkinson's Disease
Brief Title: The Effect of Repetitive Transcranial Magnetic Stimulation on Cognitive Impairment in Parkinson's Disease (PD)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Asmaa Hasan, Asmaa Mohamed Mohamed Mahmoud Hasan Assistant Lecturer of Neurology, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: rTMS and cognition in PD
Record Dates: First submitted 2019-03-14; First posted 2019-03-18 (Actual); Last update posted 2021-12-21 (Actual); Status verified 2020-07

CONDITIONS: Parkinson's Disease With Cognitive Impairment
MeSH Terms: interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Real rTMS (Active Comparator): Real rTMS high frequency stimulation (25 HZ), with intensity of 80% of resting motor threshold detected from the hand motor area, with total 2000 pulses for each hemisphere on the hand motor area for 10 consecutive sessions totally over period of 10 days.
  Interventions: Device: repetitive Transcranial Magnetic Stimulation
- Sham rTMS (Sham Comparator): Sham rTMS high frequency stimulation (25 HZ), with intensity of 80% of resting motor threshold detected from the hand motor area, with total 2000 pulses for each hemisphere with coil perpendicular on scalp for 10 consecutive sessions totally over period of 10 days.
  Interventions: Device: repetitive Transcranial Magnetic Stimulation

INTERVENTIONS:
Device: repetitive Transcranial Magnetic Stimulation — By defining intensity of 80% of the resting Motor Threshold detected from motor area for Rt Abductor digiti minimi (ADM), we will apply repetitive Transcranial Magnetic Stimulation (rTMS) using 70-mm diameter air-cooled figure-of-8 coil and SuperRapid2 Magnetic Stimulator with high frequency (25Hz), Stimuli will be delivered for total 2000 pulse (divided on 50 trains with 40 pulses per train with inter-train interval 30 seconds) for each hemisphere (coil placed tangential over the optimal position of hand motor area detected for Real group and the same coil placed perpendicular with hand of coil pointing upward over occipital cortex for Sham group). Sessions will be consecutive for ten days period with repetition of consecutive 5 sessions as boosting doses on 5 days period over the follow up visits every month for the next 3 months.
  Other Names: rTMS

SUMMARY:
This study aims to assess the therapeutic role of rTMS on parkinson's patients with cognitive impairment. Patients diagnosed with Parkinson's Disease and cognitive impairment will be recruited. All patients will be admitted and will be allocated randomly into two groups one of which will receive real sessions of high frequency rTMS for each hemisphere for 10 consecutive sessions totally over period of 10 days with repeated booster sessions every month during the period of follow up. The other will receive sham sessions.

DETAILED DESCRIPTION:
This study aims to assess the therapeutic role of rTMS on parkinson's patients with cognitive impairment. Thirty PD patients with cognitive impairment using United Kingdom (UK ) bank criteria for PD will be recruited from outpatient clinic in Assiut University. All patients will be admitted at Neuropsychiatric Department, Assiut University Hospital/ Assiut, Egypt.Each patient fulfilled the inclusion criteria as having score less than 24 on Mini-Mental Status Examination will be recruited. The patients will be allocated randomly into two groups one of which will receive real sessions of high frequency rTMS (25 HZ), with intensity of 80% of resting motor threshold detected from the hand motor area, with total 2000 pulses for each hemisphere for 10 consecutive sessions totally over period of 10 days with repeated booster session every month during the period of follow up among three months. The other will receive sham sessions. All subjects will be followed up by selected clinical rating scales at different intervals pre session, post 10 sessions, and after one, two and three months.

ELIGIBILITY:
Inclusion Criteria:

* All patients with Parkinson's Disease who were diagnosed according to UK bank criteria for PD, Aged 45-75 years, with criteria for cognitive impairment (Mini-Mental Status Examination< 24), and consent obtained from the patient or his caregiver.

Exclusion Criteria:

* History of repeated head injury
* History of repeated cerebrovascular strokes
* History of defined encephalitis
* Oculogyric crisis, supranuclear gaze palsy
* Family history of more than one relative
* History of drug intake as antipsychotics or 1-methyl-4-phenyl-1,2,3,6-tetrahydropyridine (MPTP) exposure
* Moderate and Severe depression (Hamilton Depression Rating Scale score >16)
* severe dysautonomia
* Cerebellar signs
* Babinski sign
* Strictly unilateral features after 3 years
* Hydrocephalus or intracranial lesion on neuroimaging
* We also excludes patients with intracranial metallic devices or with pacemakers or any other device.

Ages: 45 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2019-03-15 (Actual); Primary Completion 2019-06-15 (Actual); Study Completion 2019-06-15 (Actual)

PRIMARY OUTCOMES:
changes in Mini Mental State Examination (MMSE) | three months
  any changes in MMSE along the course of follow up (baseline, post treatment, one, two and three months later). Any score greater than or equal to 24 points (out of 30) indicates a normal cognition. Below this, scores can indicate severe (≤9 points), moderate (10-18 points) or mild (19-23 points) cognitive impairment.
changes in Montreal cognitive assessment scale (MoCA) | 3 months
  any changes of Montreal cognitive assessment scale (MoCA)along the course of follow up (baseline, post treatment, one, two and three months later). MoCA scores range between 0 and 30. A score of 26 or over is considered to be normal. In a study, people without cognitive impairment scored an average of 27.4; people with mild cognitive impairment (MCI) scored an average of 22.1; people with Alzheimer's disease scored an average of 16.2.
Event related potential P300 | 10 days
  changes in Event related potential P300 latency and amplitude (pre sessions -post sessions)As cognitive impairment elongates the P300 latency, we hypotheses that P300 could be a monitoring biomarker for rTMS effect, on cognitive function.

SECONDARY OUTCOMES:
motor part of Unified Parkinson's disease rating scale (UPDRS) | 3 months
  changes in motor part of Unified Parkinson's disease rating scale (UPDRS)along the course of follow up (baseline, post treatment, one, two and three months later)
changes in cortical excitability | 10 days
  changes in cortical excitability (baseline, post treatment)

CONTACTS AND LOCATIONS:
Overall Officials: Eman Khedr, Professor, Study Director — Neurology Department, Faculty of Medicine, Assiut University
Locations (1):
- Assiut University, Asyut, Egypt

REFERENCES:
- [Background] Aarsland D, Andersen K, Larsen JP, Lolk A, Kragh-Sorensen P. Prevalence and characteristics of dementia in Parkinson disease: an 8-year prospective study. Arch Neurol. 2003 Mar;60(3):387-92. doi: 10.1001/archneur.60.3.387. PMID 12633150
- [Background] Aarsland D, Bronnick K, Fladby T. Mild cognitive impairment in Parkinson's disease. Curr Neurol Neurosci Rep. 2011 Aug;11(4):371-8. doi: 10.1007/s11910-011-0203-1. PMID 21487730
- [Background] Aarsland D, Ballard C, Rongve A, Broadstock M, Svenningsson P. Clinical trials of dementia with Lewy bodies and Parkinson's disease dementia. Curr Neurol Neurosci Rep. 2012 Oct;12(5):492-501. doi: 10.1007/s11910-012-0290-7. PMID 22806065
- [Background] Chaudhuri KR, Prieto-Jurcynska C, Naidu Y, Mitra T, Frades-Payo B, Tluk S, Ruessmann A, Odin P, Macphee G, Stocchi F, Ondo W, Sethi K, Schapira AH, Martinez Castrillo JC, Martinez-Martin P. The nondeclaration of nonmotor symptoms of Parkinson's disease to health care professionals: an international study using the nonmotor symptoms questionnaire. Mov Disord. 2010 Apr 30;25(6):704-9. doi: 10.1002/mds.22868. PMID 20437539
- [Derived] Khedr EM, Mohamed KO, Ali AM, Hasan AM. The effect of repetitive transcranial magnetic stimulation on cognitive impairment in Parkinson's disease with dementia: Pilot study. Restor Neurol Neurosci. 2020;38(1):55-66. doi: 10.3233/RNN-190956. PMID 31815705